CLINICAL TRIAL: NCT00270543
Title: A Phase II Study of Bi-Weekly Docetaxel Plus 24-Hour Infusion of High-Dose 5-Fluorouracil and Leucovorin(HDFL)for Inoperable Advanced or Metastatic Gastric Cancer
Brief Title: An Effective and Well-Tolerated Regimen of Docetaxel Plus High-Dose 5-Fluorouracil and Leucovorin(HDFL)to Treat Inoperable Advanced or Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-93006
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2004-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Taxotere, Fluorouracil, Leucovorin

SUMMARY:
The primary endpoint of this phase II trial is the objective tumor response rate. The secondary endpoints include treatment-related toxicity, the clinical benefit response defined by the change in performance status and body weight, the change in quality of life, progression free survival and overall survival. Simon's optimal two-stage design will be used to determine the patient number.

DETAILED DESCRIPTION:
The regimen consists of docetaxel, 50 mg/m2, 5-FU, 2400 mg/m2, and leucovorin, 240 mg/m2 on days 1 and 15. Docetaxel will be given by 1-hour intravenous infusion and 5-FU/leucovorin by 24-hour intravenous infusion.

The treatment cycle will be repeated every 4 weeks. Dexamethasone will be given before and after each docetaxel infusion to prevent hypersensitivity and fluid retention. Tumor response will be evaluated every 2 cycles. For patients with inoperable locally advanced disease on entry, those who achieve clinical complete (CR) and partial (PR) response will be evaluated for the feasibility of curative surgical resection.If pathological CR is documented, at least 2 cycles of chemotherapy will be given after surgery. If microscopic residual tumor is noted after curative surgery, protocol treatment will be continued until disease progresses or intolerable toxicities develop. For patients with metastatic diseases on entry, those who achieve CR will receive at least 2 more cycles of chemotherapy after documentation of CR. Patients with PR will continue protocol treatment until disease progresses or intolerable toxicities develop. Patients with stable disease will continue protocol treatment if there are minor tumor responses or improvement of their general condition; patients will stop protocol treatment and change to salvage therapy if no any clinical benefits are observed. Patients with progressive disease should stop protocol treatment and change to salvage therapy.

The primary endpoint of this phase II trial is the objective tumor response rate. The secondary endpoints include treatment-related toxicity, the clinical benefit response defined by the change in performance status and body weight, the change in quality of life, progression free survival and overall survival. Simon's optimal two-stage design will be used to determine the patient number.If 5 or more objective responses are documented in the first 19 patients, the study will go on to the second stage to enroll a total of 54 eligible patients. The P0, P1,are 20%, 40%, 0.05, and 0.1, respectively. Assuming a dropout rate of 10%, 21 patients will be accrued in the first stage and 39 in the second stage. Estimated time for patient accrual is 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically proven and inoperable advanced gastric adenocarcinoma. 2.Bi-dimensionally measurable disease by physical examination or image study (roentgenogram or computed tomography scan). The index lesions should be at least 20 mm × 10 mm in size. 3.Age must be older than 18 and younger than 75 year-old. 4.Karnofsky performance status 60%. 5.Adequate bone marrow reserves, defined as white blood cell (WBC) 4,000/l, absolute neutrophil count (ANC)1,500/l, platelet 100,000/l. 6.Liver transaminases 2.5 times upper normal limit if no liver metastasis and 5 times upper normal limit if liver metastasis is present; total bilirubin 1.5 mg/dl; serum creatinine 1.5 mg/dl. 7.Serum triglyceride level 70 mg/dl. 8.Previous chemotherapy for metastatic disease is not allowed in this study. Previous adjuvant chemotherapy following curative gastrectomy is acceptable if the adjuvant chemotherapy has been completed for more than 6 months before enrollment into the present study. 9.Previous radiotherapy is allowed if the treatment was completed at least 4 weeks before the enrollment into this study. 10.Patients of childbearing age should have effective contraception during the study period. 11.All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

* 1.Patients who are receiving concurrent radiotherapy, chemotherapy or other experimental therapy. 2.Patients who refuse port-A catheter implantation. 3.Patients with brain or leptomeningeal metastases. 4.Patients who have significant cardiac arrhythmia or acute myocardial infarction within 6 months before entry. 5.Patients who have major systemic diseases that the attending physicians considered inappropriate for systemic chemotherapy. 6.Life expectancy less than 2 months. 7.Pregnant or nursing women may not participate. Women or men with reproductive potential may not participate unless they have agreed to use an effective contraceptive method. 8.No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancers, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any cancer from which the patient has been disease-free for 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine the tumor response rate of bi-weekly docetaxel plus 24-hour infusion of
high-dose 5-FU/leucovorin chemotherapy for patients with inoperable advanced gastric cancer.

SECONDARY OUTCOMES:
The rate of clinical benefit response defined by improvement in at least one of the 2 parameters
performance status and weight gain.
Toxicities of bi-weekly docetaxel plus 24-hour infusion of high-dose 5-FU/leucovorin chemotherapy
The patients'quality of life as evaluated by questionnaire interview Time to disease progression
Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Huei Yeh, Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Kun-Huei Yeh, Taipei, Ban-Ciao, Taiwan